CLINICAL TRIAL: NCT04540835
Title: Evaluation of the Effectiveness of Calcium-Phosphate-Containing Desensitizing Agent on Postoperative Sensitivity in Composite Restorations: A Double-Blind Prospective Randomized Controlled Study
Brief Title: Evaluation of the Effectiveness of Calcium Phosphate Containing Desensitizer on Postoperative Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Leyla Kerimova, Principal Investigator, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: DKA20/15
Record Dates: First submitted 2020-08-27; First posted 2020-09-07 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Teethmate (Experimental): Half of the cavities will be applied Teethmate Desensitizer following manufacturer instructions before restoration
  Interventions: Device: Teethmate Desensitizer (Kuraray)
- Negative Control (No Intervention): Half of the cavities will be restored without application of Teethmate Desensitizer

INTERVENTIONS:
Device: Teethmate Desensitizer (Kuraray) — Calcium phosphate desensitizer applied after caries removal. After restored using an oblique incremental technique with a composite resin (Filtek Z250, 3M Espe, USA)
  Arms: Teethmate

SUMMARY:
In this randomized clinical study, we aim to evaluate the effects of Teethmate Desensitizer on postoperative sensitivity when applied underneath the composite restoration by comparing it with the negative control group.

DETAILED DESCRIPTION:
For the purpose of statistical preliminary analysis, the part related to the comparison of the dependent two sample means (t test) was used in the G * power 3.1 program. The power of the test was taken as 90%, margin of error 5% and effect size 0.50. The total sample size was found to be 44. In this study, the required number of participants was determined to be at least 44, since the split-mouth technique in which both the experimental and the control groups will be used in each patient, and the number of participants to be included in the study was determined as 50 considering the ''drop-outs'' that may occur during the study. Then, randomization will be achieved using the blocked randomization technique. Randomization will be done on www.sealedenvelope.com website. For blocked randomization, the seed number will be 12345 and the block width will be 2.

After applying to Başkent University Faculty of Dentistry, dental caries are detected as a result of the clinical and radiological examination, and female or male patients will be selected among the ones who are referred to the Restorative Dentistry Department's clinic for treatment. Participation in the study is on a voluntary basis and the participants who accept the invitation will have the Informed Consent Form read and signed. If deemed necessary, the participants will be given oral hygiene motivation and initiatives will be started after their oral hygiene is achieved to a satisfactory level.

Before starting treatment of individuals diagnosed with caries clinically and radiologically, the vitality of the relevant teeth will be measured using a vitalometer (Model D624, Parkell Inc, USA). After the opening of 2 cavities in each participant, the cavities will be isolated, and Teethmate Desensitizer will be applied randomly to one of the two cavities. In order to ensure randomization, the randomization list prepared using the program on www.sealedenvelop.com will be put in an opaque envelope. When the application will be made, the envelope will be opened. Then, CaOH(Dycal, Dentsply, USA) will be placed in the deepest place where the pulp is closest. Restorations will be performed after the matrix system is applied when necessary. All cavities one-step self-etch an adhesive (Clearfil SE Bond, Kuraray Noritake, Tokyo, Japan) LED light applied according to the user instructions (Ledmax Cordless 550 Benlioğlu, Turkey)> 1,500mw / cm2 for 10 seconds polymerized. The teeth will be restored using an oblique incremental technique with a composite resin (Filtek Z250, 3M Espe, USA). Each layer will be polymerized for 20 sec. Finishing and polishing process will be done using diamond finishing burs, tires and polishing discs (Soflex, 3M Espe, USA). Restoration will be done by a single operator (LK). After the restoration, patients will be given two forms, one for each tooth, where they will record their daily pain levels for a week, and how to register on this form will be explained. These forms given to the participants will include a Numerical Rating Scale (NRS) with scores between 0-4 and a Visual Analogue Scale (VAS) of 0-100mm for 1 week. When patients will be called to the control appointment after a week, the forms in which they score the sensitivity level will be taken back. 6 weeks after the restorations are applied, the patients will be invited to a control appointment and the restorations will be checked. At the first week and sixth week control appointments, the restorations will be evaluated by another physician (KY). At the end of the 6 week, the vitality will be controlled. During the six-week study, patients will be asked not to use any pain medication, and if the participant uses painkillers during the study, the participant will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Accepting to participate
2. Being in the age range of 18-65
3. Presence of at least 12 teeth in occlusion
4. The teeth to be included in the study have natural opposite and aproximal teeth
5. The teeth to be included in the study will be vital
6. The anterior or posterior teeth to be included in the study, regardless of the deep carious cavity type, have a primary carious lesion that is estimated to be very close to the pulp during cavity preparation but the pulp will not expose (dentin thickness close to the remaining pulp is less than 2 mm)
7. In the patient's mouth, one on the right and the other on the left 4., 5. and 6. 2 teeth matching the criteria.

Exclusion Criteria:

* Not accepting voluntarily to participate in the study 2- Being younger than 18 years old or over 65 years old 3- Presence of spontaneous toothache or orofacial pain 4- Bruxism 5- Presence of advanced periodontal disease 6- The presence of a serious systemic disease. 7- Worn, cracked or devital teeth with enough material loss to be crowned 8- Presence of lesions in the apical region after radiographic examination 9- Exposure of pulp during cavity preparation 10- Presence of gingival recession 11- Individuals who have taken painkillers, anti-inflammatory and psychotropics in the last two weeks and are currently taking 12- Pregnancy and breastfeeding individuals 13- Individuals who are allergic to the materials to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kerimova, DDS, Principal Investigator — Baskent University School of Dentistry
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: restorations
Groups:
- All Study Participants: Since the study was designed as split-mouth, each participant had 2 restorations (experimental and control group) .
  The study groups allocated according to randomisation list created in www.sealedenvelope.com
Period: Week 1
Arm/Group | All Study Participants
Started | 50; 100 restorations (Participants between 18-51 years-old, and the average age was 30 years.)
Teethmate Desensitizer | 49; 49 restorations
Negative Control | 49; 49 restorations
Completed | 49; 98 restorations
Not Completed | 1; 2 restorations
Not completed — Lost to Follow-up | 1
Period: Week 6
Arm/Group | All Study Participants
Started | 49; 98 restorations (Male 14, female 33 completed the 6-week study as one subject was excluded from the study because of a newly learned pregnancy, and one refused to continue because of severe hypersensitivity in a tooth with no TD pretreatment.)
Teethmate Desensitizer | 47; 47 restorations
Negative Control | 47; 47 restorations
Completed | 47; 94 restorations
Not Completed | 2; 4 restorations
Not completed — Pregnancy | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis included participants whose treated teeth responded positively to the electric pulp test. Each participant was examined intraorally using an electric pulp tester, and only teeth that responded to the vitality test were considered vital and included in the study.
Units Other Than Participants: teeth
Groups:
- Experimental (Teethmate) and Control Groups: Since the study was designed as split-mouth, all participants had both experimental and control groups .
Arm/Group | Experimental (Teethmate) and Control Groups
Number analyzed (Participants) | 50
Number analyzed (teeth) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (12)
Sex/Gender, Customized [Number; unit: participants] — Population: overall 50 participants enrolled
  participants
    All genders | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Preoperative Vitality Measurement [Count of Units; unit: teeth] — Pulp vitality of each tooth was evaluated using a D624 pulp tester (Parkell Inc, Edgewood, NY, USA.). A toothpaste was applied to the probe tip, and the electrode was placed on the middle third of the buccal surface. The device intensity was gradually increased until the participant felt a mild tingling sensation. If the patient feels an uncomfortable sensation, such as tingling, warmth, or pain, the tooth pulp is considered vital. No score recording was performed. Electric pulp tester used only for checking the vitality of teeth and excluding them in case of negative (nonvital) response.
  teeth | 100

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: Postoperative hypersensitivity was evaluated using a 10-cm Visual Analogue Scale (VAS). The scale consisted of a straight 10-cm line with endpoints defining extreme limits: "no pain at all" (score = 0) and "pain as bad as it could be" (score = 10). Participants were asked to mark their perceived pain level on the line between the two endpoints. The distance (in cm) from the "no pain" end to the mark represented the participant's pain score. Higher scores indicated greater hypersensitivity (worse outcome).
Time Frame: 7 days after restoration
Measure: Mean (Standard Deviation); unit: cm on a 10-point Visual Analogue Scale
Units Other Than Participants: restorations
Groups:
- Teethmate: Half of the cavities will be applied Teethmate Desensitizer following manufacturer instructions before restoration
  Teethmate Desensitizer (Kuraray): Calcium phosphate desensitizer applied after caries removal. After restored using an oblique incremental technique with a composite resin (Filtek Z250, 3M Espe, USA) POS after 6 weeks was reported in 34% of teeth of experimental group.
- Negative Control: Half of the cavities will be restored without application of Teethmate Desensitizer.
  POS after 6 weeks was reported in 40.4% of teeth of control group.
Arm/Group | Teethmate | Negative Control
Number analyzed (Participants) | 49 | 49
Number analyzed (restorations) | 49 | 49
cm on a 10-point Visual Analogue Scale | 0.4 (1.6) | 1.3 (5.1)

2. Primary Outcome: Numerical Rating Scale (NRS)
Description: Progress of postoperative hypersensitivity will be also evaluated by using Numerical Rating Scale with five possibilities for the patient to state how much sensitivity there is in each tooth. The patients will have the option of saying whether the sensitivity was equal to 0 (none), 1 (mild), 2 (moderate), 3 (considerable), or 4 (severe). The mean and standard deviation (SD) of NRS scores were calculated for each group.
Time Frame: 7 days after restoration
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: restorations
Arm/Group | Teethmate | Negative Control
Number analyzed (Participants) | 49 | 49
Number analyzed (restorations) | 49 | 49
score on a scale | 0.1 (0.3) | 0.1 (0.3)

3. Secondary Outcome: Presence of Postoperative Hypersensitivity (Patient-reported at 6 Weeks)
Description: This patient-reported outcome was pre-specified in the study protocol to assess the presence of postoperative hypersensitivity at 6 weeks.
Time Frame: 6 weeks after restoration
Measure: Count of Units; unit: restorations
Units Other Than Participants: restorations
Arm/Group | Teethmate | Negative Control
Number analyzed (Participants) | 47 | 47
Number analyzed (restorations) | 47 | 47
restorations | 47 | 47

ADVERSE EVENTS:
Time Frame: Up to 7 days and 6 weeks after restorative procedure
Description: Participants were actively and systematically monitored for any adverse events, including temporary sensitivity, discomfort, or soft tissue irritation, during treatment and at follow-up visits after the restorative procedures.
  Of the 50 total participants, 49 attended the 1-week and 47 attended the 6-week follow-up. No non-serious adverse events were reported or observed during the study period.
Groups:
- All Participants: Because this was a split-mouth design, each participant received both interventions (Teethmate and Control) on different teeth. Therefore, adverse events could not be attributed to a single intervention. Adverse event data are reported for all participants combined.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04540835/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT04540835/ICF_001.pdf